CLINICAL TRIAL: NCT04110145
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Sequential, Ascending, Multidose Study to Evaluate the Safety and Efficacy of Linaclotide in Pediatric Participants (Age 2 to 5 Years) With Functional Constipation
Brief Title: Linaclotide Safety and Efficacy in 2 to 5-Year-Old Participants With Functional Constipation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Collaborators: Ironwood Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: LIN-MD-67; 2019-002126-75 (EudraCT Number)
Record Dates: First submitted 2019-09-27; First posted 2019-10-01 (Actual); Results first posted 2022-04-26 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-03

CONDITIONS: Functional Constipation
Keywords: Functional constipation in children; LINZESS
MeSH Terms: interventions — linaclotide

STUDY DESIGN:
Intervention Model Description: There are 3 cohorts with ascending doses and an additional final cohort to repeat the highest dose determined to be safe
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1 (Linaclotide 18 μg) (Experimental): Linaclotide 18 microgram (μg), capsules, mixed with water and administered orally, once daily in fasted state (30 minutes before any meal) for the 4-week Study Intervention Period.
  Interventions: Drug: Linaclotide
- Cohort 2 (Linaclotide 36 μg) (Experimental): Linaclotide 36 μg, capsules, mixed with water and administered orally, once daily in fasted state (30 minutes before any meal) for the 4-week Study Intervention Period.
  Interventions: Drug: Linaclotide
- Cohort 3 (Linaclotide 72 μg) (Experimental): Linaclotide 72 μg, capsules, mixed with water and administered orally, once daily in fasted state (30 minutes before any meal) for the 4-week Study Intervention Period.
  Interventions: Drug: Linaclotide
- Final Cohort (Linaclotide 72 μg) (Experimental): Linaclotide at the highest dose tested/determined to be safe (72 μg), capsules, mixed with water and administered orally, once daily in fasted state (30 minutes before any meal) for the 4-week Study Intervention Period.
  Interventions: Drug: Linaclotide
- Placebo Pooled (Placebo Comparator): Matching placebo, orally, once daily in fasted state (30 minutes before any meal) for the 4-week Study Intervention Period pooled from Cohorts 1, 2, 3, and Final Cohort.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Linaclotide — Linaclotide, capsules, mixed with water and administered orally, once daily in fasted state.
  Arms: Cohort 1 (Linaclotide 18 μg); Cohort 2 (Linaclotide 36 μg); Cohort 3 (Linaclotide 72 μg); Final Cohort (Linaclotide 72 μg)
Drug: Placebo — Matching placebo, capsules, mixed with water and administered orally, once daily in fasted state
  Arms: Placebo Pooled

SUMMARY:
The purpose of this study is to evaluate the dose response, safety, and efficacy of linaclotide when compared with placebo in pediatric participants, 2 to 5 years of age, with Functional Constipation.

ELIGIBILITY:
Inclusion Criteria:

* Participant weighs ≥10 kilograms (kg) at the time the parent/guardian/legally authorized representative (LAR) has provided signed consent
* Participant meets modified Rome III criteria for FC: For at least 2 months before Screening (Visit 1) (for participants aged ≥ 4 years old), or for at least 1 month before Screening (Visit 1) (for participants aged < 4 years old), the participant has had 2 or fewer defecations (with each defecation occurring in the absence of any laxative, suppository, or enema use during the preceding 24 hours) per week.

In addition, at least once per week, participant must meet 1 or more of the following:

1. History of retentive posturing or excessive volitional stool retention
2. History of painful or hard bowel movements (BMs)
3. Presence of a large fecal mass in the rectum
4. History of large diameter stools that may obstruct the toilet
5. At least one episode of fecal incontinence per week after the acquisition of toileting skills

   * Participant is willing to discontinue any laxatives used before the Preintervention Visit in favor of the protocol-permitted rescue medicine
   * Parent/guardian/LAR and caregiver must provide written informed consent before the initiation of any study-specific procedures
   * Caregiver who will be completing the eDiary is able to read and/or understand the assessments in the eDiary device and must undergo training

Exclusion Criteria:

* For participants aged ≥ 4 years old: Participant meets Rome III criteria for Child/Adolescent IBS: At least once per week for at least 2 months before Screening (Visit 1), the participant has experienced abdominal discomfort (an uncomfortable sensation not described as pain) or pain associated with 2 or more of the following at least 25% of the time:

  1. Improvement with defecation
  2. Onset associated with a change in frequency of stool
  3. Onset associated with a change in form (appearance) of stool
* Participant has required manual dis-impaction any time prior to randomization or dis-impaction during in-patient hospitalization within 1 year prior to randomization
* Participant currently has both unexplained and clinically significant alarm symptoms (lower GI bleeding [rectal bleeding or heme-positive stool], iron-deficiency anemia, or any unexplained anemia, or weight loss) and systemic signs of infection or colitis, or any neoplastic process
* Participant has had surgery that meets any of the following criteria:

  1. Surgery to remove a segment of the GI tract at any time before Screening (Visit 1)
  2. Surgery of the abdomen, pelvis, or retroperitoneal structures during the 6 months before the Screening Visit
  3. An appendectomy or cholecystectomy during the 60 days before Screening (Visit 1)
  4. Other major surgery during the 30 days before Screening (Visit 1)
* Participant has a mechanical bowel obstruction or pseudo-obstruction.
* Participant has a known allergy or sensitivity to the study intervention or its components or other medications in the same drug class
* Participant has any of the following conditions:

  1. Celiac disease, or positive serological test for celiac disease or the condition is suspected but has not been ruled out by endoscopic biopsy
  2. Cystic fibrosis
  3. Hypothyroidism that is untreated or treated with thyroid hormone at a dose that has not been stable for at least 3 months prior to Screening (Visit 1)
  4. Down's syndrome or any other chromosomal disorder
  5. Active anal fissure (ie, participant reports having streaks of blood on the stool or on toilet paper and/or pain/crying with bowel movement within 2 weeks prior to Screening). (Note: Anal fissures that have resolved at least 2 weeks prior to screening would not be exclusionary.) However, if in the investigator's opinion, an anal fissure(s) may be the primary cause of participant's modified Rome III FC criteria, the participant would not be eligible to participate in the study.
  6. Anatomic malformations (eg, imperforate anus, anal stenosis, anterior displaced anus)
  7. Intestinal nerve or muscle disorders (eg, Hirschprung disease, visceral myopathies, visceral neuropathies)
  8. Neuropathic conditions (eg, spinal cord abnormalities, neurofibromatosis, tethered cord, spinal cord trauma)
  9. Lead toxicity, hypercalcemia
  10. Neurodevelopmental disabilities (early-onset, chronic disorders that share the essential feature of a predominant disturbance in the acquisition of cognitive, motor, language, or social skills, which has a significant and continuing impact on the developmental progress of an individual) producing a cognitive delay that precludes comprehension and completion of the daily eDiary or other study-related questionnaires (Note: Participants are excluded if the person who will be completing the daily eDiary or other study-related questionnaires meets this criterion.)
  11. Inflammatory bowel disease
  12. Childhood functional abdominal pain syndrome
  13. Childhood functional abdominal pain
  14. Poorly treated or poorly controlled psychiatric disorders that might influence his or her ability to participate in the study
  15. Lactose intolerance that is associated with symptoms which could confound the assessments in this study
  16. History of cancer other than treated basal cell carcinoma of the skin. (Note:

Participants with a history of cancer are allowed provided that the malignancy has been in a complete remission before the Randomization Visit. A complete remission is defined as the disappearance of all signs of cancer in response to treatment.)

* Participant received a study intervention during the 30 days before Screening (Visit 1) or is planning to receive study intervention (other than that administered during this study)
* Participant's parent/guardian/LAR or caregiver has been directly or indirectly involved in the conduct and administration of this study as an investigator, study coordinator, or other study staff member. In addition, any participant, parent/guardian/LAR or caregiver who has a first-degree family member, significant other, or relative residing with him/her directly or indirectly who is involved in this study
* For participants aged ≥ 4 years old: Participant has a history of non-retentive fecal incontinence

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2021-04-20 (Actual); Study Completion 2021-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Muslin, Study Director — Allergan
Locations (18):
- United States (18):
  - Central Research Associates, Inc, Birmingham, Alabama
  - HealthStar Research, Hot Springs, Arkansas
  - Preferred Clinical Research Partners, Little Rock, Arkansas
  - Advanced Research Center, Anaheim, California
  - Kindred Medical Institute for Clinical Trials, LLC, Corona, California
  - Center for Clinical Trials, LLC, Paramount, California
  - Prohealth Research Center, Doral, Florida
  - South Miami Medical & Research Group, Inc., Miami, Florida
  - River Birch Research Alliance, LLC, Blue Ridge, Georgia
  - SleepCare Research Institute, Inc., Stockbridge, Georgia
  - Virgo Carter Pediatrics, Silver Spring, Maryland
  - Minnesota Gastroenterology PA, Minneapolis, Minnesota
  - David M. Headley, MD, P.A., Port Gibson, Mississippi
  - Foundation Pediatrics Med Clinical Research Partners, LLC, East Orange, New Jersey
  - Advantage Clinical Trials, The Bronx, New York
  - Coastal Pediatric Research, Charleston, South Carolina
  - Coastal Pediatric Research, Mt. Pleasant, South Carolina
  - Clinical Research Partners, LLC, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Allergan will share de-identified patient-level data and study-level data including protocols and clinical study reports for phase 2 - 4 trials completed after 2008 that are registered to ClinicalTrials.gov or EudraCT, have received regulatory approval in the United States and/or the European Union in a given indication and the primary manuscript from the trial has been published. To request access to the data, the researcher must sign a data use agreement and any shared data is to be used for non-commercial purposes. More information can be found on http://www.allerganclinicaltrials.com/.
Supporting Information: Study Protocol, CSR
Time Frame: After having received regulatory approval in the United States and/or the European Union in a given indication and the primary manuscript from the trial has been published.
Access Criteria: To request access to the data, the researcher must sign a data use agreement and any shared data is to be used for non-commercial purposes.
URL: http://www.allerganclinicaltrials.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized in a 3:1 ratio to receive ascending doses of linaclotide Cohorts 1-3 (18/36/72 μg) to determine the highest dose to be safe or placebo and in a 5:1 ratio for the Final Cohort (72 μg) safe dose or placebo.
Period: Double-Blind Treatment Period (4 Weeks)
Arm/Group | Cohort 1 (Linaclotide 18 μg) | Cohort 2 (Linaclotide 36 μg) | Cohort 3 (Linaclotide 72 μg) | Final Cohort (Linaclotide 72 μg) | Placebo Pooled
Started | 7 | 7 | 6 | 7 | 8
Completed (Completed= Participants who completed the Double-Blind Treatment Period) | 7 | 7 | 6 | 6 | 8
Not Completed | 0 | 0 | 0 | 1 | 0
Not completed — Site Terminated by the Sponsor | 0 | 0 | 0 | 1 | 0
Period: Post-Treatment Period (1 Week)
Arm/Group | Cohort 1 (Linaclotide 18 μg) | Cohort 2 (Linaclotide 36 μg) | Cohort 3 (Linaclotide 72 μg) | Final Cohort (Linaclotide 72 μg) | Placebo Pooled
Started (Started=Participants who entered the Post-Treatment Period) | 7 | 7 | 5 | 6 | 8
Completed | 7 | 7 | 5 | 6 | 8
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Modified Intent-to-Treat Population (mITT) included all Randomized Population who received at least 1 dose of double-blind study intervention and who had at least 1 postbaseline entry on bowel movement (BM) characteristic assessments that determine occurrences of spontaneous bowel movements (SBMs).
Groups:
- Cohort 1 (Linaclotide 18 μg): Linaclotide,18 μg, capsules, orally, once daily in fasted state (30 minutes before any meal) for the 4-week Study Intervention Period.
- Cohort 2 (Linaclotide 36 μg): Linaclotide, 36 μg, capsules, orally, once daily in fasted state (30 minutes before any meal) for the 4-week Study Intervention Period.
- Cohort 3 (Linaclotide 72 μg): Linaclotide, 72 μg, capsules, orally, once daily in fasted state (30 minutes before any meal) for the 4-week Study Intervention Period.
- Final Cohort (Linaclotide 72 μg): Linaclotide at the highest dose tested/determined to be safe (72 μg), capsules, orally, once daily in fasted state (30 minutes before any meal) for the 4-week Study Intervention Period.
- Placebo Pooled: Matching placebo once daily in fasted state (30 minutes before any meal) for the 4-week Study Intervention Period pooled from Cohorts 1, 2, 3, and Final Cohort.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (Linaclotide 18 μg) | Cohort 2 (Linaclotide 36 μg) | Cohort 3 (Linaclotide 72 μg) | Final Cohort (Linaclotide 72 μg) | Placebo Pooled | Total
Number analyzed (Participants) | 7 | 7 | 6 | 7 | 8 | 35
Age, Continuous [Mean (Full Range); unit: years] | 3.6 [2 to 5] | 3.3 [2 to 5] | 4.0 [3 to 5] | 3.6 [2 to 5] | 3.5 [3 to 4] | 3.6 [2 to 5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 5 | 0 | 4 | 16
  Male | 3 | 4 | 1 | 7 | 4 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 4 | 4 | 3 | 14
  Not Hispanic or Latino | 6 | 5 | 2 | 3 | 5 | 21
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 4 | 2 | 2 | 3 | 16
  White | 2 | 3 | 4 | 5 | 5 | 19
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in 4-week Overall Spontaneous Bowel Movement (SBM) Frequency Rate (SBMs/Week) During the Study Intervention Period of Each Cohort
Description: A SBM was defined as a bowel movement (BM) that occurred in the absence of laxative, suppository, or enema use on the calendar day of the BM or the calendar day before the BM. Each day the caregiver recorded the number of SBMs in the last 24 hours in an electronic diary (eDiary). The SBM frequency rate (SBMs/week) during the analysis period for each participant was calculated as [(total number of SBMs in the analysis period/number of days in the analysis period)*7]. Baseline value was based on values collected 14 days before randomization up to randomization. Change from Baseline was calculated as the SBM frequency rate during the 4-week treatment period - SBM frequency rate at Baseline. A positive change from Baseline indicates improvement.
Time Frame: Baseline (14 days prior to randomization) to Day 29
Population: mITT Population included all Randomized Population who received at least 1 dose of double-blind study intervention and who had at least 1 postbaseline entry on BM characteristic assessments that determine occurrences of SBMs.
Measure: Mean (Standard Deviation); unit: SBMs per week
Arm/Group | Cohort 1 (Linaclotide 18 μg) | Cohort 2 (Linaclotide 36 μg) | Cohort 3 (Linaclotide 72 μg) | Final Cohort (Linaclotide 72 μg) | Placebo Pooled
Number analyzed (Participants) | 7 | 7 | 6 | 7 | 8
SBMs per week
  Baseline | 1.379 (1.095) | 0.621 (0.365) | 0.724 (0.953) | 1.034 (0.809) | 1.267 (1.062)
  Change from Baseline to Day 29 | 3.100 (5.251) | 0.032 (0.508) | 3.603 (2.867) | 1.574 (1.933) | 0.482 (0.773)

2. Primary Outcome: Change From Baseline in 4-week Stool Consistency Reported by the Caregiver During the Study Intervention Period of Each Cohort
Description: The caregiver rated and recorded in an eDiary the consistency of the stool for each bowel movement using the Bristol Stool Form 7-point scale where: 1=Separate hard lumps, like nuts (hard to pass); 2=Sausage-shaped, but lumpy; 3=Like a sausage but with cracks on its surface; 4=Like a sausage or snake, smooth and soft; 5=Soft blobs with clear cut edges (easy to pass); 6=Fluffy pieces with ragged edges, a mushy stool; 7=Watery, no solid pieces. Entirely liquid. Baseline value was based on values collected 14 days before randomization up to randomization. A participant's stool consistency score for the treatment period was the average of the nonmissing consistency scores from the BMs recorded by the caregiver during the 4-week treatment period.
Time Frame: Baseline (14 days prior to randomization) to Day 29
Population: mITT Population included all Randomized Population who received at least 1 dose of double-blind study intervention and who had at least 1 postbaseline entry on BM characteristic assessments that determine occurrences of SBMs. Overall number analyzed are the number of participants with data available for analyses.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 1 (Linaclotide 18 μg) | Cohort 2 (Linaclotide 36 μg) | Cohort 3 (Linaclotide 72 μg) | Final Cohort (Linaclotide 72 μg) | Placebo Pooled
Number analyzed (Participants) | 5 | 5 | 3 | 7 | 7
score on a scale
  Baseline | 1.633 (0.461) | 1.700 (0.447) | 2.733 (1.079) | 2.021 (0.793) | 2.024 (0.641)
  Change from Baseline to Day 29 | 0.917 (1.360) | 1.600 (1.294) | 1.687 (2.779) | 1.716 (1.689) | 0.596 (0.937)

3. Primary Outcome: Change From Baseline in 4-week Straining Reported by the Caregiver During the Study Intervention Period of Each Cohort
Description: The caregiver rated and recorded in an eDiary the amount of straining they observed when the child passed the BM (1=Not at all; 2=Yes a little; 3=Yes a lot; I don't know). Baseline value was based on values collected 14 days before randomization up to randomization. A participant's straining score for the treatment period was the average of the nonmissing straining scores from the BMs recorded by the caregiver during the 4-week treatment period. A negative change from Baseline indicates improvement.
Time Frame: Baseline (14 days prior to randomization) to Day 29
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: straining score
Arm/Group | Cohort 1 (Linaclotide 18 μg) | Cohort 2 (Linaclotide 36 μg) | Cohort 3 (Linaclotide 72 μg) | Final Cohort (Linaclotide 72 μg) | Placebo Pooled
Number analyzed (Participants) | 5 | 5 | 3 | 7 | 7
straining score
  Baseline | 2.310 (0.410) | 2.600 (0.379) | 2.600 (0.361) | 2.571 (0.426) | 2.548 (0.658)
  Change from Baseline to Day 29 | -0.370 (0.631) | -0.320 (0.325) | -0.769 (0.884) | -0.996 (0.759) | -0.334 (0.360)

4. Primary Outcome: Percentage of Days With Fecal Incontinence During the Study Intervention Period (for Participants Who Have Acquired Toileting Skills During the Daytime and Nighttime or Acquired Toileting Skills During Daytime Only) Within Each Cohort
Description: Each day the caregiver recorded in an eDiary if the child had a bowel movement accident (Yes; No; I don't know). The percentage of days with fecal incontinence for the treatment period was the average of the nonmissing incidences of fecal incontinence recorded by the caregiver during the 4-week treatment period.
Time Frame: 29 Days
Population: mITT Population included all Randomized Population who received at least 1 dose of double-blind study intervention and who had at least 1 postbaseline entry on BM characteristic assessments that determine occurrences of SBMs. Number analyzed is the number of participants with data available for analyses.
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Cohort 1 (Linaclotide 18 μg) | Cohort 2 (Linaclotide 36 μg) | Cohort 3 (Linaclotide 72 μg) | Final Cohort (Linaclotide 72 μg) | Placebo Pooled
Number analyzed (Participants) | 5 | 6 | 5 | 5 | 6
percentage of days | 0.007 (0.016) | 0.065 (0.107) | 0.091 (0.063) | 0.009 (0.019) | 0.000 (0.000)

5. Primary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: An Adverse Event (AE) is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease. A Serious Adverse Event (SAE) is defined as any untoward medical occurrence that: results in death, is immediately life-threatening, requires in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, and/or causes a congenital anomaly/birth defect. A TEAE is an AE that begins or worsens after receiving study drug. Safety Population included all participants in the Randomized Population who received at least 1 dose of double-blind study intervention.
Time Frame: First dose of study drug intervention to within 1 week of last dose (Up to 45 days)
Population: Safety Population included all participants in the Randomized Population who received at least 1 dose of double-blind study intervention.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1 (Linaclotide 18 μg) | Cohort 2 (Linaclotide 36 μg) | Cohort 3 (Linaclotide 72 μg) | Final Cohort (Linaclotide 72 μg) | Placebo Pooled
Number analyzed (Participants) | 7 | 7 | 6 | 7 | 8
percentage of participants
  TEAEs | 28.6 | 0.0 | 0.0 | 28.6 | 12.5
  TESAE | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

ADVERSE EVENTS:
Time Frame: First dose of study drug intervention to within 1 week of last dose (Up to 45 days)
Description: All-Cause Mortality: All randomized participants. Serious Adverse Events and Other Adverse Events: Safety Population included all participants in the Randomized Population who received at least 1 dose of double-blind study intervention.
Arm/Group | Cohort 1 (Linaclotide 18 μg) | Cohort 2 (Linaclotide 36 μg) | Cohort 3 (Linaclotide 72 μg) | Final Cohort (Linaclotide 72 μg) | Placebo Pooled
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7 | 0/6 | 0/7 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 0/6 | 0/7 | 0/8
Other Adverse Events (participants affected / at risk) | 2/7 | 0/7 | 0/6 | 2/7 | 1/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (Linaclotide 18 μg) (N=7) | Cohort 2 (Linaclotide 36 μg) (N=7) | Cohort 3 (Linaclotide 72 μg) (N=6) | Final Cohort (Linaclotide 72 μg) (N=7) | Placebo Pooled (N=8)
Otitis media (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Developmental delay (General disorders) | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2020-05-04): https://cdn.clinicaltrials.gov/large-docs/45/NCT04110145/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-11): https://cdn.clinicaltrials.gov/large-docs/45/NCT04110145/SAP_001.pdf